CLINICAL TRIAL: NCT06870747
Title: Application of Ultra Low Frequency TENS During Non-surgical Periodontal Treatment Relieves Pain and Discomfor
Brief Title: Use of TENS in Non-surgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Sara Di Nicolantonio, Professor, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UL'Aquila
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-01

CONDITIONS: Non-surgical Periodontal Therapy
Keywords: ULF-TENS; pain; non-surgical periodontal therapy; scaling
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): patients who undergo non-surgical periodontal therapy with TENS switch on
  Interventions: Device: use of Transcutaneous electrical neurostimulation
- Control group (Active Comparator): patients who undergo non-surgical periodontal therapy with TENS switch off
  Interventions: Device: no TENS during non-surgical periodontal therapy

INTERVENTIONS:
Device: use of Transcutaneous electrical neurostimulation — in this study we would like to use for the first time TENS device during non surgical periodontal therapy
  Arms: Experimental group
Device: no TENS during non-surgical periodontal therapy — patients in the control group are going to have non surgical periodontal therapy without TENS
  Arms: Control group

SUMMARY:
the aim of the study is to verify the use of TENS in non-surgical periodontal therapy in order to relief pain

DETAILED DESCRIPTION:
non-surgical periodontal therapy could be painfull for some patients and the pain that they may experience can let them avoid therapies, with huge risks for their oral health. Transcutaneous electrical neurostimulation (TENS) is a device largely used in temporomandibular disorders in order to reduce pain. The aim of our study is to analyze the effect of Transcutaneous electrical neurostimulation (TENS) at the tragus during non-surgical periodontal therapy fro pain relief

ELIGIBILITY:
Inclusion Criteria:

* Patients aging more than 18 and of both sexes seeking for non-surgical periodontal treatment

Exclusion Criteria:

* Patients following opioids or analgesic therapies during the study

  * Pregnant women
  * Patients who have had episodes of epilepsy
  * Pace-maker patients
  * Patients who did not signed the informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Tooth pain during non surgical periodontal therapy | 30 minutes
  we are going to measure pain with VAS scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, L’Aquila, Aquila, Italy

IPD SHARING:
Plan to Share IPD: No